CLINICAL TRIAL: NCT04926454
Title: Effect of Dexmedetomidine as an Adjuvant to Bupivacaine in Ultrasound Guided Transversus Abdominis Plane Block Versus Caudal Block for Post-operative Analgesia in Children Undergoing Congenital Inguinal Hernia Repair
Brief Title: Efficacy of Adding Dexmedetomidine as an Adjuvant to Bupivacaine in TAP Block and Caudal Block
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU M S 484 / 2020
Record Dates: First submitted 2021-05-23; First posted 2021-06-15 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Experimental): patients will receive general anesthesia followed by Tap block at the end of the operation.
  Interventions: Drug: Dexmedetomidine
- Caudal block (Experimental): patients will receive general anesthesia followed by caudal block at the beginning of the operation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will be monitored using standard monitoring (heart rate, non-invasive blood pressure, ECG and pulse oximetery) After the child is adequately anesthetized, intra-venous access with appropriate size cannula will be obtained Appropriate size LMA (2 and 2.5) will be inserted and patients will be allowed to breathe spontaneously.
  patients will receive 0.25% Bupivacaine (0.3ml/Kg) with 1 μg/kg dexmedetomidine After general anaesthesia
  Other Names: Bupivacaine

SUMMARY:
This study compares the efficacy of Dexmedetomidine as an adjuvant to Bupivacaine in Ultrasound Guided Transversus Abdominis Plane Block versus Caudal Block for post-operative analgesia in children undergoing congenital inguinal hernia repair especially to provide prolonged post-operative analgesia and decrease opioid consumption.

DETAILED DESCRIPTION:
Inguinal hernia is the most common lower abdominal surgery of childhood. It results from a small sac that comes through the inguinal ring that is normally open during fetal life and closes around the time of birth. For reasons we don't understand, it does not close in some infants. This sac then makes a pathway for abdominal organs to come through the inguinal ring into the groin . In boys, the organ is usually a loop of bowel and in girls; it may be bowel or an ovary. In boys and girls, the hernia first appears as a bulge in the groin. It usually "pops out" when the child cries or strains. If only fluid comes through the inguinal ring into the sac, the problem is called a hydrocele. It is treated via a low transverse incision to repair the defect.

Postoperatively, patients experience somatosensory pain from the incision site and visceral irritation and discomfort .

The impact of painful experience on the young nervous system is so significant that long-term effects can occur, including a lowered pain tolerance for months after a pain-producing event however, the benefits of adequate analgesia include attenuation of the surgical stress response, decreased perioperative morbidity and improved outcome in certain types of surgery. Also effective pain control facilitates rehabilitation and accelerates recovery from surgery .

Regional anesthesia and analgesia techniques are commonly used to facilitate pain control during pediatric surgical practice, decrease parenteral opioids requirements and improve the quality of post-operative pain control and patient-parent satisfaction.

Caudal epidural anesthesia is considered the gold standard regional technique for pain management after pediatric pelvic and lower abdominal procedures because it blocks both somatic and visceral pain. The caudal block has a low complication rate (0.7 per 1000) , provides 4 to 6 hours of analgesia, and results in improved patient pain scores than in patients having general anesthesia alone .

An increased understanding of abdominal wall anatomy has led to the introduction of the transversus abdominis plane block (TAPB) for managing pain after lower abdominal surgery .TAPB provides reliable unilateral sensory block in the T10-L1 distribution with a single injection, and resulted in a significant decrease in postoperative pain scores and opioid requirements after major abdominal surgeries . Similar outcomes have been observed in pediatric studies, and analgesia after TAPB in pediatric patients is thought to last 10 to 15 hours .

The technique of TAP block has been found to be a safe and effective tool in a variety of general, gynaecological, and urological surgery, and it is suggested as part of the multimodal anaesthetic approach to enhance recovery after lower abdominal surgeries .

However, the duration of analgesia provided by these strategies is limited by the short duration of action of the local anesthetic .

Various adjuvants to local anesthetics have been investigated to improve the quality of block and duration of analgesia, including Dexmedetomidine, fentanyl, morphine, ketamine, midazolam, and magnesium.

Each of these adjuvants has side effects specific to the type and dose of adjuvant used. For instance, behavioral changes have been noted with the use of caudal ketamine, opioids are associated with risk of respiratory depression, and the neurotoxicity of midazolam is still controversial. Therefore, an ideal adjuvant that provides maximal analgesia with minimal side effects for these blocks is still a matter of contention.

Dexmedetomidine (DEX) is a highly selective α2-adrenoceptor agonist, possesses sedative, analgesic, anxiolytic, and anti-inflammatory properties . When administered in combination with local anesthetics in the epidural space, it has been shown to reduce postoperative analgesic requirements and have a significantly

ELIGIBILITY:
Inclusion Criteria:

* age 2-12 years
* Elective congenital inguinal hernia repair operation under general anaesthesia.
* Physical Status: ASA I and II Patients after taking written and informed consent from the parents or care giver.

Exclusion Criteria:

* Refusal of procedure or participation in the study by parents.
* Physical status: ASA III or above.
* Children undergoing bilateral lower abdominal surgeries.
* Infection at site of injection.
* Congenital anomaly of the spine.
* History of developmental delay, neurological disease, skeletal deformities.
* History or evidence of coagulopathy.
* Allergies to drugs used (Bupivacaine 0.5%)( dexmedetomidine/prcedex)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-10-25 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
When Dexmedetomidine is administered in combination with local anesthetics in the epidural space, it has been shown to reduce postoperative analgesic requirements and have a significantly analgesic effect" | Within 24 hours post operative
  The primary outcome measures were the time to first analgesia (in minutes from the time of caudal (or) TAP block injection to first registration of modified VAS scale ≥3 at any point of time will receive paracetamol 10mg/kg orally

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Eldeen Ewis, Professor, Study Chair — Professor of Anesthesia, intensive care and pain management
Locations (1):
- AinShams Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis — https://pubmed.ncbi.nlm.nih.gov/23811424/
- See also: Effect of adding dexamethasone to bupivacaine on transversus abdominis plane block for abdominal hysterectomy: A prospective randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/23162395/
- See also: Cutaneous flexion reflex in human neonates: a quantitative study of threshold and stimulus-response characteristics after single and repeated stimuli — https://pubmed.ncbi.nlm.nih.gov/10587047/
- See also: Assessment and management of inguinal hernia in infants — https://pubmed.ncbi.nlm.nih.gov/23008462/
- See also: Effect of low dose dexmedetomidine premedication on propofol consumption in geriatric end stage renal disease patients — https://pubmed.ncbi.nlm.nih.gov/26323728/
- See also: Intraoperative dexmedetomidine attenuates postoperative systemic inflammatory response syndrome in patients who underwent percutaneous nephrolithotomy: a retrospective cohort study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5818878/
- See also: Caudal anesthesia in pediatrics: an update — https://pubmed.ncbi.nlm.nih.gov/16682915/
- See also: Analgesic effect of perineural magnesium sulphate for sciatic nerve block for diabetic toe amputation: A randomized trial — https://pubmed.ncbi.nlm.nih.gov/28464014/
- See also: Applications of regional anaesthesia in paediatrics — https://pubmed.ncbi.nlm.nih.gov/24335395/
- See also: Comparison of Dexmedetomidine and Fentanyl as an Adjuvant to Ropivacaine for Postoperative Epidural Analgesia in Pediatric Orthopedic Surgery — https://pubmed.ncbi.nlm.nih.gov/28332374/
- See also: Analgesia Following Arthroscopy - a Comparison of Intra-articular Bupivacaine and/or Midazolam and or Fentanyl — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5339352/
- See also: Transversus abdominis plane block in children: a multicenter safety analysis of 1994 cases from the PRAN (Pediatric Regional Anesthesia Network) database — https://pubmed.ncbi.nlm.nih.gov/24918899/
- See also: Epidemiology and morbidity of regional anaesthesia in children — https://pubmed.ncbi.nlm.nih.gov/18458552/
- See also: Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/22632762/